CLINICAL TRIAL: NCT03717181
Title: Expanded Access Use of Lixivaptan in a Single Subject With Intractable Pain Due to Polycystic Kidney Disease
Brief Title: Lixivaptan in a Single Subject With Intractable Pain Due to Polycystic Kidney Disease
Status: No longer available | Type: Expanded Access
Sponsor: Palladio Biosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: PA-103
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: Polycystic Kidney
MeSH Terms: conditions — Polycystic Kidney Diseases | interventions — lixivaptan

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Lixivaptan — Daily dose of lixivaptan optimized using a predetermined titration protocol.

SUMMARY:
Abdominal pain, sometimes severe, is a known symptom of polycystic kidney disease (PKD) related to the cystic expansion. This study will investigate whether the vasopressin V2 receptor antagonist lixivaptan can alleviate intractable pain in a pediatric PKD patient who cannot tolerate the related vasopressin V2 receptor antagonist tolvaptan.

ELIGIBILITY:
Inclusion Criteria:

1. Capable of understanding the written informed consent/assent.
2. Provides signed and witnessed written informed consent/assent, and agrees to comply with protocol requirements and study-related procedures.
3. At least 15 years of age at the time of Screening.
4. Subject has been diagnosed with ADPKD by modified Ravine criteria:

   * If the subject has a family history of ADPKD, a minimum of 3 cysts per kidney by sonography or 5 cysts by computerized tomography or MRI; or
   * If the subject does not have a family history of ADPKD, a minimum of 10 cysts per kidney by any radiologic method and exclusion of other cystic kidney diseases.
5. Considered by the Investigator to be in good health relative to underlying CKD status and clinically stable with respect to underlying CKD, based on medical evaluation that includes medical and surgical history, as well as a complete physical examination including vital signs, ECG, and laboratory test results.

Exclusion Criteria:

1. Has a known sensitivity or idiosyncratic reaction to any compound present in lixivaptan or any compound listed as being present in the formulation.
2. Is pregnant or breast feeding.
3. Has taken any investigational drug or used an investigational device within 30 days or 5 half-lives, whichever is longer, prior to Screening.
4. Has taken tolvaptan, conivaptan, somatostatin analogs (e.g. lanreotide, pasireotide, octreotide, etc.), mTOR kinase inhibitors (e.g. everolimus, sirolimus, etc.), or oral or intravenous antibiotics within 30 days or 5 half-lives, whichever is longer, prior to Day 1.
5. Has a history of testing positive for hepatitis B surface antigen, hepatitis C, or human immunodeficiency virus (HIV).
6. Consumes grapefruit or Seville oranges (or their juices, or foods containing their extract) from 7 days prior to the first dose of study medication and until after the final dose.
7. Has clinically significant liver disease, or clinically significant liver function abnormalities or serology other than that expected for ADPKD with cystic liver disease at baseline.
8. Has any clinically significant laboratory abnormalities or concomitant conditions other than ADPKD (including treatment for such conditions) that, in the opinion of the Investigator, could either interfere with the study drug or pose an unacceptable risk to the subject.

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Marie C Hogan, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States